CLINICAL TRIAL: NCT03476941
Title: Antibiotic Irrigations for Intra-Abdominal Drains
Acronym: AID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Paolo Goffredo (Other)
Responsible Party: Sponsor-Investigator, Paolo Goffredo, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201703759
Record Dates: First submitted 2017-08-09; First posted 2018-03-26 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Abdominal Abscess
MeSH Terms: conditions — Abdominal Abscess | interventions — Injections; clindamycin phosphate

STUDY DESIGN:
Intervention Model Description: There will be two group, study and control group. In control group, patient will receive standard intra-abdominal drain care with daily flushing of the drain with normal saline. In study group, patient will receive daily flush with antibiotic for 7 days.
Who Masked: Participant
Masking Description: Written consent will be obtained from all participants. Then, each participant will be randomized into two arms. Nurse will administer the drain flush either with normal saline or antibiotic irrigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Antibiotic Irrigation (Experimental): The drain will be irrigated twice/day with the above antibiotic solution for 7 days maximum
  Interventions: Drug: Gentamicin Sulfate Inj 20mg/2ml vial for injection; Drug: Clindamycin phosphate 6 mg/1ml for injection
- Normal Saline Irrigation (Placebo Comparator): The drain will be irrigated twice/day with normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gentamicin Sulfate Inj 20mg/2ml vial for injection — Irrigate surgical drain with total amount of 5 mg in 10 ml volume twice/day for 7 days or until drain removal if less than 7 days of therapy.
  Arms: Antibiotic Irrigation
Drug: Clindamycin phosphate 6 mg/1ml for injection — Irrigate surgical drain with total amount of 12 mg in 10 ml volume once daily for 7 days or until drain removal if less than 7 days of therapy.
  Arms: Antibiotic Irrigation
Other: Placebo — The placebo group will receive drain irrigation twice/day
  Arms: Normal Saline Irrigation

SUMMARY:
Intra-abdominal abscesses are pus-filled pouches in the abdominal cavity. Current standard of care includes drain placement in the abscess cavity to reach source control as well as administration of systemic antibiotics. It is common practice to flush the drain on a daily basis to ensure patency. This study aims to analyze the clinical impact of a higher local concentration of antibiotics (rather than normal saline) provided through drain irrigation with an antimicrobial agent (Gentamicin and/or Clindamycin) compare to normal saline.

DETAILED DESCRIPTION:
People with an abdominal abscess who undergo drain placement will have those drains irrigated twice/day with either normal saline (placebo group) or with the above antibiotic solution for a total of 7 days or less if the drain were to be removed earlier. Outcomes of interest are duration of systemic antibiotics, and WBC and temperature curve.

ELIGIBILITY:
Inclusion Criteria:

* Intra-abdominal abscess drained with catheter/drain
* Treatment with systemic antibiotics
* Able to consent

Exclusion Criteria:

* Abscess(es) not amendable for an image guided drain placement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Duration of systemic antibiotics | From initiation of systemic treatment until 1 month follow up
  Total duration of systemic antibiotics will be recorded from the start of the treatment until discontinuation by primary care team. This will be measured as days from diagnosis to when the antibiotic treatment gets interrupted. Duration of systemic antibiotics will be our primary outcome measurement. Duration of systemic antibiotics will be monitored as an indication of the effectiveness of the proposed intervention.

SECONDARY OUTCOMES:
White Blood Count | From initiation of systemic treatment until 1 month follow up
  White blood count level from the blood draw will be measured starting from the admission until discharge or discontinuation by primary care team. During follow up, if white blood count will be measured, will record up to 1 month follow up. The white blood count will be measured once daily and as needed depending on clinical changes. We will plan to trend WBC as another indication of decreasing systemic inflammation.
Change in temperature | From initiation of systemic treatment until 1 month follow up
  Temperature will be measured every 8 hours starting from admission and until patient discharge. And also temperature will be measured during each follow up clinic visit. Change in temperature is monitored as an indication of decrease systemic inflammation.
Changes in size of the Abscess | From patient initial hospitalization up to 1 month follow up
  CT scan of would have been obtained prior to image guided drain placement. Any subsequent CT scans up to 1 month follow up upon discharge will be reviewed to assess changes in size of the abscess. This will be monitored for assessing the effectiveness of intervention.
Changes in Drain Output | From the drain placement up to 1 month follow up
  Drain will have certain output that is recorded daily. Daily drain output will be in unit of ml and will be monitored as a measurement of abscess resolution.
Duration of drain | From the drain placement until 1 month follow up
  The total duration of the drain placement will be recorded in days starting from the day of placement up to drain removal and monitored as a effectiveness of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Goffredo, MD, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
At this point, there is no IPD sharing plan and not included in the consent process.

REFERENCES:
- [Background] Yoon YI, Hwang S, Cho YJ, Ha TY, Song GW, Jung DH. Therapeutic effect of trans-drain administration of antibiotics in patients showing intractable pancreatic leak-associated pus drainage after pancreaticoduodenectomy. Korean J Hepatobiliary Pancreat Surg. 2015 Feb;19(1):17-24. doi: 10.14701/kjhbps.2015.19.1.17. Epub 2015 Feb 28. PMID 26155272
- [Background] Sauermann R, Karch R, Kjellsson MC, Feurstein T, Puspok A, Langenberger H, Bohmdorfer M, Jager W, Zeitlinger M. Good penetration of moxifloxacin into human abscesses. Pharmacology. 2012;90(3-4):146-50. doi: 10.1159/000341550. Epub 2012 Aug 3. PMID 22868236
- [Background] Sauermann R, Feurstein T, Karch R, Kjellsson MC, Jager W, Bohmdorfer M, Puspok A, Langenberger H, Wild T, Winkler S, Zeitlinger M. Abscess penetration of cefpirome: concentrations and simulated pharmacokinetic profiles in pus. Eur J Clin Pharmacol. 2012 Oct;68(10):1419-23. doi: 10.1007/s00228-012-1270-1. Epub 2012 Mar 23. PMID 22441316
- [Background] Zimmerman LH, Tyburski JG, Glowniak J, Singla R, Lavery T, Nailor M, Stassinopoulus J, Hong K, Barshikar S, Dolman HS, Baylor AE, Wilson RF. Impact of evaluating antibiotic concentrations in abdominal abscesses percutaneously drained. Am J Surg. 2011 Mar;201(3):348-52; discussion 352. doi: 10.1016/j.amjsurg.2010.09.010. PMID 21367377